CLINICAL TRIAL: NCT07153770
Title: Bozitinib Combined With Chemotherapy as Radical Treatment for Stage IIA-IIIC MET-Altered Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Chunxia Su, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025LY0214
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: NSCLC; MET Exon 14 Mutation; MET Activating Mutation
Keywords: NSCLC; Bozitinib; Radical Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bozitinib group (Experimental): Participants will receive bozitinib in combination with standard platinum-based doublet chemotherapy for 8 weeks. Following investigator-assessed operability, surgical resection will be performed approximately 4 weeks after completion of neoadjuvant therapy. The first MRD assessment will be conducted after completion of neoadjuvant therapy and before surgery.A second MRD assessment will be performed within 7 days to 1 month after surgery. Based on a comprehensive evaluation of MRD status, tumor markers, and imaging results, if molecular abnormalities are detected., patients will receive bozitinib within 3 months after surgery. If CEA remains within the normal range and blood cfDNA-MRD is negative, patients will enter a regular follow-up program, with MRD assessments every 3 months during the first 2 years and every 6 months from years 3 to 5. If MRD conversion to positive, abnormal CEA, or abnormal CT findings occur within 5 within 5 years, bozitinib will be administered.
  Interventions: Drug: Bozitinib

INTERVENTIONS:
Drug: Bozitinib — Participants will receive bozitinib in combination with standard platinum-based doublet chemotherapy for 8 weeks. Following investigator-assessed operability, surgical resection will be performed approximately 4 weeks after completion of neoadjuvant therapy. The first MRD assessment will be conducted after completion of neoadjuvant therapy and before surgery.A second MRD assessment will be performed within 7 days to 1 month after surgery. Based on a comprehensive evaluation of MRD status, tumor markers, and imaging results, if molecular abnormalities are detected., patients will receive bozitinib within 3 months after surgery. If CEA remains within the normal range and blood cfDNA-MRD is negative, patients will enter a regular follow-up program, with MRD assessments every 3 months during the first 2 years and every 6 months from years 3 to 5. If MRD conversion to positive, abnormal CEA, or abnormal CT findings occur within 5 within 5 years, bozitinib will be administered.

SUMMARY:
This study aim to evaluate the efficacy and safety of Bozitinib combined with chemotherapy as radical treatment for stage IIA-IIIC MET-altered non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria to participate in this study:
* Signed informed consent.
* Age ≥ 18 years.
* Histologically or cytologically confirmed NSCLC adenocarcinoma, with -postoperative pathology confirming stage IIA-IIIC.
* Willing to undergo curative resection, and assessed by a surgeon as operable with no surgical contraindications.
* No prior systemic anti-tumor therapy.
* Expected survival ≥ 6 months.
* At least one measurable or evaluable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0-2.
* MET alteration confirmed by NGS gene testing, including the following types:

MET exon 14 skipping mutation (NGS results from tissue or blood sample certified by CLIA or CAP).

* MET primary amplification, NGS positive or FISH GCN ≥6 (results from tissue or blood sample certified by CLIA or CAP or FISH assay).
* MET protein overexpression, immunohistochemistry showing ≥50% tumor cells with ++ or higher staining.
* Adequate pulmonary function to tolerate surgery.
* Adequate organ and bone marrow function, defined as:
* Hematology: absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L; platelets ≥ 100 × 10⁹/L; hemoglobin ≥ 9.0 g/dL.
* Hepatic function: total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); for patients with HCC, liver metastases, or history/suspected Gilbert syndrome (persistent or recurrent hyperbilirubinemia, mainly unconjugated, without evidence of hemolysis or liver lesions), TBIL ≤ 3 × ULN; for patients without HCC or liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN.
* Renal function: serum creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance (CCr) ≥ 50 mL/min; urine dipstick protein < 2+.
* Coagulation: activated partial thromboplastin time (APTT) and international normalized ratio (INR) ≤ 1.5 × ULN.

Thyroid function: normal thyroid-stimulating hormone (TSH); if baseline TSH is outside the normal range, enrollment is allowed if total T3 (or FT3) and FT4 are within normal limits.

* Cardiac enzymes: within normal range (isolated laboratory abnormalities deemed clinically insignificant by the investigator are acceptable).
* Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 3 days prior to the first dose of study drug (Cycle 1, Day 1). If urine pregnancy test cannot be confirmed negative, a serum pregnancy test is required. Non-childbearing females are defined as postmenopausal for at least 1 year, or surgically sterile (bilateral oophorectomy or hysterectomy).

All subjects with potential risk of pregnancy (male or female) must use highly effective contraception with a failure rate <1% during treatment and for 120 days after the last dose of study drug (or 180 days after the last dose of chemotherapy).

Exclusion Criteria:

* Patients meeting any of the following criteria are not eligible for this study:

Presence of EGFR, ALK, ROS1, or other actionable mutations excluding MET. Receipt of live attenuated vaccines within 4 weeks prior to enrollment or planned during the study period.

* All participants must undergo brain imaging (MRI or contrast-enhanced CT) prior to enrollment to rule out brain metastases.
* Major surgery (e.g., thoracic, abdominal, or pelvic) within 4 weeks prior to study treatment initiation, or ongoing recovery from surgical complications.

Diagnosis of any malignancy other than NSCLC within 5 years prior to study treatment initiation (excluding completely resected basal cell carcinoma or squamous cell carcinoma of the skin, in situ carcinoma, or completely resected papillary thyroid carcinoma).

* Active, known, or suspected autoimmune disease.
* Known history of primary immunodeficiency.
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* Known hypersensitivity to the study drug bozitinib, platinum-based doublet chemotherapy, or any excipients.
* Not fully recovered from any toxicity and/or complications caused by prior interventions (i.e., ≤ Grade 1 or returned to baseline, excluding fatigue or alopecia) prior to study treatment.
* Untreated active hepatitis B infection (defined as HBsAg positive with detectable HBV-DNA above the upper limit of normal at the local laboratory).

Note: Patients with hepatitis B meeting the following criteria may be enrolled:

HBV viral load <1000 copies/mL (200 IU/mL) prior to first dose; patients must receive antiviral therapy throughout chemotherapy to prevent viral reactivation.

Patients who are anti-HBc (+), HBsAg (-), anti-HBs (-), and HBV viral load (-) do not require prophylactic antiviral therapy but must be closely monitored for viral reactivation.

* Active hepatitis C infection (HCV antibody positive and HCV-RNA above the assay lower limit of detection).
* Any history, condition, treatment, or laboratory abnormality that could interfere with study results, hinder full participation, or that the investigator considers a potential risk or inappropriate for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2027-09-20 (Estimated); Study Completion 2028-09-20 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response | Up to 6 month
  defined as the proportion of patients who achieve a major pathological response among all patients undergoing surgical pathological assessment. Major pathological response is defined as ≤10% viable tumor cells in the resected primary tumor and regional lymph nodes, as assessed by hematoxylin and eosin (H&E) staining.

SECONDARY OUTCOMES:
Objective Response Rate | Up to 6 month
  defined as the proportion of patients who achieve a complete response (CR) or partial response (PR) among all patients.
Pathological Complete Response rate | Up to 6 month
  defined as the proportion of patients who achieve a pathological complete response among all patients undergoing surgical pathological assessment. Pathological complete response is defined as the absence of any residual viable tumor cells in the resected primary tumor and regional lymph nodes, as assessed by hematoxylin and eosin (H&E) staining.
Disease Control Rate | Up to 2 year
  defined as the proportion of patients who achieve stable disease (SD), partial response (PR), or complete response (CR) among all patients.
Event-Free Survival | Up to 2 year
  defined as the time from randomization to disease progression precluding surgery, local or distant disease recurrence, or death from any cause, whichever occurs first.
3-Year Overall Survival | Up to 3 year
  defined as the proportion of patients who are alive within 3 years from the time of randomization among all patients.
Overall Survival | Up to 5 year
  defined as the time from randomization to death from any cause.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code